CLINICAL TRIAL: NCT03584633
Title: Standardization of Indocyanine Green Lymphography Protocol With Exercise for Lymphedema Assessment
Brief Title: Effect of Exercise on Indocyanine Green (ICG) Lymphography Imaging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201803867
Record Dates: First submitted 2018-06-05; First posted 2018-07-12 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lymphedema
Keywords: Indocyanine Green; Indocyanine Green Lymphography; Exercise
MeSH Terms: conditions — Lymphedema; Motor Activity | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lymphedema (Other): The subjects with lymphedema will be exercising on a Nu-Step exercise machine that will exercise their arms and legs simultaneously for five-minute intervals. Every five minutes their limbs will be imaged with Indocyanine Green Lymphography.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — The subjects will be exercising on a Nu-Step exercise machine that will exercise their arms and legs simultaneously for five-minute intervals. Every five minutes their limbs will be imaged with an ICG lymphography device to determine the plateau rate of indocyanine green dye after exercise.
  Other Names: NOVADAQ SPY Elite System Indocyanine Green Lymphography

SUMMARY:
Indocyanine Green (ICG) lymphography is a relatively new imaging technique that allows for quick visualization of superficial lymph flow in real-time, without radiation exposure. This imaging is useful for diagnosing and assessing lymphedema. ICG lymphography has a higher sensitivity and specificity than lymphoscintigraphy, the current gold standard imaging device for lymphedema. ICG lymphography precisely and reliably diagnoses, tracks, and stages lymphedema severity, ranging from subclinical or early lymphedema to more advanced cases. The ICG contrast dye used to visualize the lymphatic system takes approximately six hours to plateau. Therefore, patients must wait six hours between their initial and delayed scans.

The purpose of this study is to determine if exercising on a Nu-step device between ICG initial and delayed scans would shorten the period of time a patient had to spend at the hospital on the day of their ICG lymphography.

The general procedures for this involve (after selecting subjects, consenting subjects, educating the subject on the protocol, along with other appropriate measures):

* Taking baseline vitals (HR & SpO2) and limb circumference measurements
* 5-minute period of time to acquaint subject with the exercise equipment (Nu-Step) at any level of exertion
* injection of contrast agent to allow for visualization of the superficial lymphatic system by a qualified nurse
* Initial scan
* A 5-minute period of exercise at "moderate" level of exercise (This correlates to the rating of perceived exertion levels of 12-13; All exercise periods should be at this level and will be monitored by a provider)
* Second scan & vitals
* 5-minute period of exercise
* Third scan & vitals

  o Continue 5-minute exercise period followed by scan & vitals until disease pattern emerges

  * Exercise for 5 minutes then scan and vitals until images reach steady state for two consecutive scans
* Final vitals (HR & SpO2)

  * Repeat scan every 1 hour until the normal 6 hour scan to monitor for further changes in lymphatic pattern.
* Exit survey

DETAILED DESCRIPTION:
Following consent, the patients will answer the questions in the screening questionnaire and this data will be collected. Patients that do not screen out of the study (i.e. meet all inclusion criteria and none of the exclusion criteria) will continue with the study. Individuals who meet the exclusion criteria will not continue.

Study participants will be asked to go to the Rehabilitation Therapies clinic on the lower level of the main hospital for a one time visit. The visit will take approximately three to six hours.

During the visit, height and weight will be measured. Circumference measurements of the arms and legs will also be measured with a measuring tape. Bioimpedance analysis of the limb will be performed to assess the fluid content in the limbs.

Pain Ease numbing spray will have been applied to three injection sites on the affected arm or leg. 0.1ml of 0.25% Indocyanine green (ICG) dye will then be injected into the distal arm or leg at three separate sites: two interdigital injections and one injection in the volar wrist or posterior to the medial malleolus.

An immediate scan will be acquired using an ICG lymphography device. The scan will take approximately five minutes to complete. The data from this image will be considered baseline. This image is part of the patient's normal care at our institution and would be done even if the subject was not in this study.

The participant will then use the Nu-Step exercise machine for five minutes at a rate of perceived exertion (RPE) of 12-13. Heart rate will be monitored during the exercise with a pulse oximeter. After five minutes, a delayed scan will be performed with the NOVADAQ SPY Elite System and data will be recorded. The participant will continue to exercise for five minutes at an RPE of 12-13 and be scanned after every five minutes until the scans show no change in lymph pattern after two consecutive scans. The patient will be undergoing scanning and be exercising for a maximum of one hour.

Limb circumference measurements and bioimpedance scans will be repeated after exercise has been completed. The scan will be repeated every 1 hour until the normal 6-hour scan to monitor for further changes in the lymphatic pattern.

A post-intervention questionnaire will then be provided to the participant to complete discussing their exercise experience that day during the study, their previous ICG experiences, and their preference between this protocol and the current scanning process.

During the study, the subject will be told when he/she is being photographed/recorded. The injections and scans are clinically-indicated and would occur whether the individual was in the study or not. The initial and last scans are clinically indicated to determine disease status. 3) clarify how the follow-up survey is completed via email

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Suspected lymphedema or previously diagnosed lymphedema
* Between the ages of 18-85 years old.

Exclusion Criteria:

* Allergies to iodine
* pregnant
* nursing
* On daily heart medication
* Have medical conditions affecting the heart, lungs or joint conditions that prevent prolonged physical activity of the arms or legs.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei F Chen, MD, FACS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dylke ES, Schembri GP, Bailey DL, Bailey E, Ward LC, Refshauge K, Beith J, Black D, Kilbreath SL. Diagnosis of upper limb lymphedema: development of an evidence-based approach. Acta Oncol. 2016 Dec;55(12):1477-1483. doi: 10.1080/0284186X.2016.1191668. Epub 2016 Jun 22. PMID 27333213
- [Background] Lee BB, Laredo J. Contemporary role of lymphoscintigraphy: we can no longer afford to ignore! Phlebology. 2011 Aug;26(5):177-8. doi: 10.1258/phleb.2011.011e01. No abstract available. PMID 21791706
- [Background] Mihara M, Hara H, Araki J, Kikuchi K, Narushima M, Yamamoto T, Iida T, Yoshimatsu H, Murai N, Mitsui K, Okitsu T, Koshima I. Indocyanine green (ICG) lymphography is superior to lymphoscintigraphy for diagnostic imaging of early lymphedema of the upper limbs. PLoS One. 2012;7(6):e38182. doi: 10.1371/journal.pone.0038182. Epub 2012 Jun 4. PMID 22675520
- [Background] Chen WF, Zhao H, Yamamoto T, Hara H, Ding J. Indocyanine Green Lymphographic Evidence of Surgical Efficacy Following Microsurgical and Supermicrosurgical Lymphedema Reconstructions. J Reconstr Microsurg. 2016 Nov;32(9):688-698. doi: 10.1055/s-0036-1586254. Epub 2016 Aug 3. PMID 27487485
- [Background] Yamamoto T, Matsuda N, Doi K, Oshima A, Yoshimatsu H, Todokoro T, Ogata F, Mihara M, Narushima M, Iida T, Koshima I. The earliest finding of indocyanine green lymphography in asymptomatic limbs of lower extremity lymphedema patients secondary to cancer treatment: the modified dermal backflow stage and concept of subclinical lymphedema. Plast Reconstr Surg. 2011 Oct;128(4):314e-321e. doi: 10.1097/PRS.0b013e3182268da8. PMID 21921744
- [Background] Yamamoto T, Yoshimatsu H, Narushima M, Yamamoto N, Hayashi A, Koshima I. Indocyanine Green Lymphography Findings in Primary Leg Lymphedema. Eur J Vasc Endovasc Surg. 2015 Jan;49(1):95-102. doi: 10.1016/j.ejvs.2014.10.023. PMID 25488514
- [Background] International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema: 2013 Consensus Document of the International Society of Lymphology. Lymphology. 2013 Mar;46(1):1-11. PMID 23930436
- [Background] Johnson JH, Phipps LK. Preferred method of selecting exercise intensity in adult women. J Strength Cond Res. 2006 May;20(2):446-9. doi: 10.1519/R-17935.1. PMID 16686578
- [Background] Singh B, Disipio T, Peake J, Hayes SC. Systematic Review and Meta-Analysis of the Effects of Exercise for Those With Cancer-Related Lymphedema. Arch Phys Med Rehabil. 2016 Feb;97(2):302-315.e13. doi: 10.1016/j.apmr.2015.09.012. Epub 2015 Oct 9. PMID 26440777
- [Background] Morris C, Wonders KY. Concise review on the safety of exercise on symptoms of lymphedema. World J Clin Oncol. 2015 Aug 10;6(4):43-4. doi: 10.5306/wjco.v6.i4.43. PMID 26266100
- [Background] Desai P, Williams AG Jr, Prajapati P, Downey HF. Lymph flow in instrumented dogs varies with exercise intensity. Lymphat Res Biol. 2010 Sep;8(3):143-8. doi: 10.1089/lrb.2009.0029. PMID 20863266
- [Background] Downey HF, Durgam P, Williams AG Jr, Rajmane A, King HH, Stoll ST. Lymph flow in the thoracic duct of conscious dogs during lymphatic pump treatment, exercise, and expansion of extracellular fluid volume. Lymphat Res Biol. 2008;6(1):3-13. doi: 10.1089/lrb.2007.1017. PMID 18361766
- [Background] Cemal Y, Pusic A, Mehrara BJ. Preventative measures for lymphedema: separating fact from fiction. J Am Coll Surg. 2011 Oct;213(4):543-51. doi: 10.1016/j.jamcollsurg.2011.07.001. Epub 2011 Jul 28. No abstract available. PMID 21802319
- [Background] Unno N, Nishiyama M, Suzuki M, Yamamoto N, Inuzuka K, Sagara D, Tanaka H, Konno H. Quantitative lymph imaging for assessment of lymph function using indocyanine green fluorescence lymphography. Eur J Vasc Endovasc Surg. 2008 Aug;36(2):230-236. doi: 10.1016/j.ejvs.2008.04.013. Epub 2008 Jun 4. PMID 18534875
- [Background] Yamamoto T, Narushima M, Doi K, Oshima A, Ogata F, Mihara M, Koshima I, Mundinger GS. Characteristic indocyanine green lymphography findings in lower extremity lymphedema: the generation of a novel lymphedema severity staging system using dermal backflow patterns. Plast Reconstr Surg. 2011 May;127(5):1979-1986. doi: 10.1097/PRS.0b013e31820cf5df. PMID 21532424
- [Background] Yamamoto T, Yamamoto N, Doi K, Oshima A, Yoshimatsu H, Todokoro T, Ogata F, Mihara M, Narushima M, Iida T, Koshima I. Indocyanine green-enhanced lymphography for upper extremity lymphedema: a novel severity staging system using dermal backflow patterns. Plast Reconstr Surg. 2011 Oct;128(4):941-947. doi: 10.1097/PRS.0b013e3182268cd9. PMID 21681123
- [Background] Rockson SG, Rivera KK. Estimating the population burden of lymphedema. Ann N Y Acad Sci. 2008;1131:147-54. doi: 10.1196/annals.1413.014. PMID 18519968
- [Background] Lasinski BB, McKillip Thrift K, Squire D, Austin MK, Smith KM, Wanchai A, Green JM, Stewart BR, Cormier JN, Armer JM. A systematic review of the evidence for complete decongestive therapy in the treatment of lymphedema from 2004 to 2011. PM R. 2012 Aug;4(8):580-601. doi: 10.1016/j.pmrj.2012.05.003. PMID 22920313

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lymphedema
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lymphedema
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Age, Continuous [Median (Standard Deviation); unit: years] | 56.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Diseased limbs [Number; unit: limbs] | 23

OUTCOME MEASURES:

1. Primary Outcome: Time for Initial Disease Pattern to Appear
Description: After subjects exercise, this outcome will be measured by indocyanine green lymphography scans, a non-radioactive scan that visualizes the lymphatic system
Time Frame: ICG scan is performed every 5 minutes with the test subjects exercising until the initial disease pattern is seen. We expect initial disease pattern to appear within a minute following administration of ICG.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lymphedema
Number analyzed (Participants) | 9
seconds | 5 (1)

2. Secondary Outcome: Time to Reach Indocyanine Green Lymphography Steady State
Description: After subjects exercise, this outcome will be measured by indocyanine green lymphography, a non-radioactive scan that visualizes the lymphatic system.
Time Frame: ICG scan was performed every 5 minutes until lymphographic plateau was reached. The Lymphographic plateau is defined as having no observable changes in lymphographic patterns. We estimate all patients to reach plateau within 20 minutes.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lymphedema
Number analyzed (Participants) | 9
seconds | 11 (2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Lymphedema
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT03584633/Prot_SAP_002.pdf